CLINICAL TRIAL: NCT03584568
Title: Reappraising Intergeneration Relationships in Dementia Caregiving Through Perspective Taking
Brief Title: Reappraising Intergeneration Relationships in Dementia Caregiving
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Au May-lan Alma, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRFPTR2018
Record Dates: First submitted 2018-06-28; First posted 2018-07-12 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer Dementia
Keywords: Caregiving; Intergeneration; Reappraisal through perspective taking
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perspective Taking Reappraisal (Experimental): This arm focuses on reappraisals with perspective taking with a limited amount of basic skill building
  Interventions: Behavioral: Perspective Taking Reappraisal; Other: Basic Skill Building
- Basic Skill Building (Other): This arm focuses on basic skill building only.
  Interventions: Other: Basic Skill Building

INTERVENTIONS:
Behavioral: Perspective Taking Reappraisal — Interventions involving 1) appreciating relational insights; 2) enhancing self-awareness; 3) empathetic understanding of care-recipient; 4) integrating self-care and caring for others and 5) negotiation.
  Arms: Perspective Taking Reappraisal
Other: Basic Skill Building — These skill-building exercises are commonly used in psycho-education programs for caregivers:monitoring mood and activities, relaxation techniques and scheduling pleasant events, basic communication with the care recipient, communicating the caregivers' own needs with other family member or related persons including helpers and professional staff.

SUMMARY:
It is hypothesized that reappraising intergeneration relationships through perspective-taking will enhance the well-being of adult-child caregivers. Incorporating both psychological and social perspectives, the study makes a unique contribution to address research gaps by evaluating an integrated model of intervention for dementia caregivers. The conceptual model involves the following components: 1) relational insights; 2) self-reflection to integrate the challenges and benefits in caregiving; 3) interpersonal empathy

To test the incremental value of perspective-taking reappraisals, the study involves a two-arm randomized controlled trial of 12 weeks of intervention with two conditions: 1) Reappraisal through Perspective Taking and 2) Basic Skill Building. Telephone-administered sessions are integrated with group sessions and home visits to maximize sustainability and accessibility of the intervention. One hundred fifty-four participants will be recruited and randomized. Primary outcomes are reduced depressive symptoms and enhanced psychological well-being for the caregivers. Secondary outcomes include enhanced social support for caregivers and reduced behavioral problems in the care-recipients.

DETAILED DESCRIPTION:
The proposed study aims to address a major research gap in caregiving interventions in the context of intergeneration perspective-taking reappraisals. Adult child caregivers are part of a sandwich generation, involved in actualizing their own goals and coping with social expectations to care for their elderly parents. Dementia caregiving presents a particular challenge in life transition wherein the adult child is parenting his or her parents. With global aging, people living with dementia are rising exponentially. This presents a challenge for sustainable care in Hong Kong and also in countries where public services are developing and the demand for family and intergeneration caregiving is high due to collectivistic concerns. It is hypothesized that reappraising intergeneration relationships through perspective-taking will enhance the well-being of adult-child caregivers. Incorporating both psychological and social perspectives, the study makes a unique contribution to address research gaps by evaluating an integrated model of intervention for dementia caregivers. The conceptual model involves the following components: 1) relational insights; 2) self-reflection to integrate the challenges and benefits in caregiving; 3) interpersonal empathy.

Most caregiving psycho-education programs involve skill training including scheduling pleasant events, communicating with the care recipient and other family members. To test the incremental value of perspective-taking reappraisals, the study involves a two-arm randomized controlled trial of 12 weeks of intervention with two conditions: 1) Perspective Taking Reappraisal and 2) Basic Skill Building. Telephone-administered sessions are integrated with home visits to maximize sustainability and accessibility of the intervention. One hundred fifty-four participants will be recruited and randomized. Primary outcomes are reduced depressive symptoms and enhanced psychological well-being for the caregivers. Secondary outcomes include enhanced social support for caregivers and reduced behavioral problems in the care-recipients. Measures are obtained at baseline Weeks 1 (baseline), 6 and 12 with a follow-up at Week 24. Findings have implications for enhancing sustainable care for older adults in the wider society.

ELIGIBILITY:
Inclusion criteria are as follows

* Primary caregivers aged 20 or older and who have been caring for persons (aged 60 or above) with a physician diagnosis of Alzheimer's disease in the mild to moderate range as determined by the Clinical Dementia Rating Scale.
* Primary caregivers who have been providing unpaid care for more than 12 hours a week for at least the past three months.
* The care should involve day-to-day decision-making as well as any of the following: feeding, dressing, bathing, toileting, housework, preparing meals, medication and handling finances.
* They can be daughter/son or daughter-/son-in-law of the care recipient.

Exclusion criteria are as follows:

* signs of severe intellectual deficits
* demonstrated suicidal ideation
* exhibited evidence of psychotic disorders
* hearing/ visual impairment
* inability to read or speak Chinese/Cantonese fluently and severe.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2021-07-08 (Estimated); Study Completion 2021-07-08 (Estimated)

PRIMARY OUTCOMES:
Change in Center for Epidemiological Studies-Depression Search Results Center for Epidemiological Studies Depression | Week 1, 6, 12, 24
  20-item measure that asks caregivers to rate how often over the past week they The scale rates experienced symptoms associated with depression.. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater level of having depressive symptoms.
Change in Ryff's Psychological Well-being | Weeks 1,6, 12, 24
  The 18-version of the scale taps the six areas of psychological well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Respondents rate statements on a scale of 1 to 6, with 1 indicating strong disagreement and 6 indicating strong agreement. The range of scores is from 0 to 108. Higher scores suggest higher levels of well-being. The subscale score of each of the six areas can be calculating by summation of the three items associated with each of the area.

SECONDARY OUTCOMES:
Change in Revised Memory and Problem Checklist | Weeks 1, 6, 12 ,24
  The checklist is a 24-item caregiver-report measure provides a total score plus scores for three subscale memory-related problems, affective distress and disruptive behaviors. Scores are computed for the presence or absence of each problem first, and then for caregiver "reaction" or the extent to which caregivers were "bothered" or "distressed" by each behavior. The caregivers' reaction to each behavior, or the extent of distress experienced, were scored as follows: Reactions are assessed by asking how "upsetting" the behavior was on a Likert scale of 0 to 4 (0 = Not at all, 1= a little, 2 = moderately, 3 = very much, and 4 =extremely). Frequency of behaviors are assessed based on a Likert-scale of 0 to 4 (0 = never occurs, 1 = occurs infrequently and not in the last week, 2 = occurred 1-2 times in the last week, 3 = occurred 3-6 times in the last week, and 4 = occurs daily or more often). The range of score is from 0 to 96, higher scores suggesting greater disruption.
Change in MacArther Social Support Scales | Weeks 1,6, 12, 24
  The measure the levels of emotional and instrumental social support experienced by the caregivers. The scale consists of 12 items assesses the frequency of receipt of 3 categories of social support: emotional support, instrumental support and negative interaction involving conflict or excessive demands. The participants scored each item on a 5-point Likert Scale ranging from 0 (never) to 4 (frequently). The range of scores is from 0 to 48, with higher score indicating better social support.

CONTACTS AND LOCATIONS:
Overall Officials: Alma Au, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Applied Social Sciences, Hong Kong Polytechnic University, Hong Kong
  - Institute of Active Ageing, Kowloon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Au A, Gallagher-Thompson D, Wong MK, Leung J, Chan WC, Chan CC, Lu HJ, Lai MK, Chan K. Behavioral activation for dementia caregivers: scheduling pleasant events and enhancing communications. Clin Interv Aging. 2015 Mar 26;10:611-9. doi: 10.2147/CIA.S72348. eCollection 2015. PMID 25848237
- See also: Link to Project Info as funded by the University Grants Committee (General Research Fund) — https://cerg1.ugc.edu.hk/cergprod/scrrm00542.jsp?proj_id=15606317&old_proj_id=null&proj_title=connecting&isname=&ioname=&institution=&subject=&pages=1&year=2017&theSubmit=15606317